CLINICAL TRIAL: NCT02217527
Title: Development of a Novel Therapeutic for Smoking Cessation
Brief Title: Test of Novel Drug for Smoking Cessation
Acronym: UH3-P2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chengappa, K.N. Roy, MD (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kenneth A. Perkins, PhD., Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UH3-PRO14070319; UH3TR000958 (NIH)
Record Dates: First submitted 2014-07-24; First posted 2014-08-15 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Smoking Cessation
Keywords: crossover
MeSH Terms: conditions — Smoking Cessation | interventions — JNJ-39393406

STUDY DESIGN:
Intervention Model Description: Crossover of active JNJ vs. placebo for 2 weeks each, involving 1 week of dose run-up and 1 week of attempting to quit each day on that drug condition. A one-week washout separates these drug conditions, which are administered in counter-balanced order.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JNJ Active Drug (Experimental): 200 mg (100 mg b.i.d.) Active JNJ Drug used to assess quitting for one week, as part of crossover design. This JNJ experimental compound has NO name, just a company number.
  Interventions: Drug: Active JNJ Drug; Drug: Placebo pill
- Placebo Pill (Experimental): Placebo pill used for one week quit attempt, as part of crossover design.
  Interventions: Drug: Active JNJ Drug; Drug: Placebo pill

INTERVENTIONS:
Drug: Active JNJ Drug — 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week.
  Other Names: JNJ-39393406
Drug: Placebo pill — Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week.

SUMMARY:
The study will assess a novel active drug vs. placebo on ability to reduce smoking and aid cessation during a one-week "practice" quit period for each condition in smokers with a high interest in quitting (i.e. crossover design). Medication effects on reducing withdrawal and cognitive impairment will help assess the mechanism to support quit smoking attempts.

DETAILED DESCRIPTION:
We aim to test the proof of principal that an alpha-7 PAM drug, JNJ-39393406, promotes smoking cessation when compared to placebo. We have developed, tested, and validated an efficient Phase 2a screening procedure that optimally combines the validity of randomized clinical trials with the practicality of lab- based medication studies. Notably, it employs a within-subject, cross-over design comparing active versus placebo effects on quitting smoking to maximize statistical power without a large sample, in contrast to the large samples needed for between-groups randomized treatment conditions. Using this procedure, we will evaluate effects of JNJ-39393406 vs. placebo on short-term smoking abstinence in smokers who already have a high interest in quitting soon. We predict that, compared with placebo, JNJ-39393406 will increase days of abstinence, identifying initial evidence of efficacy for smoking cessation. Our main dependent measure is days of very stringent biochemically validated (expired CO<5 ppm) 24-hr smoking abstinence, with post-quit withdrawal and cognitive function as secondary measures. Potential for adverse side-effects will be assessed at each visit.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and female dependent smokers wanting to quit soon

-

Exclusion Criteria:

* Use of non-smoked nicotine products
* Already enrolled in cessation program.

  * Recent alcohol or substance dependence (≤ 3 months)
  * Women who are pregnant, planning a pregnancy, or lactating; all female participants shall undergo a pregnancy test at screening and will be excluded if positive.
  * Serious or unstable medical disorder within the past 3 months
* Epilepsy

  * Current diagnosis (within last 6-months) of abnormal cardiac rhythms; unstable cardiovascular disease e.g. stroke, myocardial infarction in the last 6 months
  * Evidence impaired liver function test (LFT)
  * Evidence of kidney failure
  * Any subject with a history of hematological cancers examples: leukemia, lymphoma etc.
  * Any clinically significant hematological laboratory abnormality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2017-07 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Perkins, PhD, Principal Investigator — Univ of PIttsburgh
Locations (1):
- Univ of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled after confirmation of eligibility were then assigned to Order 1 or Order 2.
Groups:
- Order 1--JNJ Active Then Plac: 200 mg (100 mg b.i.d.) Active JNJ Drug used to assess quitting for one week, as part of crossover design, followed by trying to quit for one week on placebo. This JNJ experimental compound has NO name, just a company number.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week.
  Placebo pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week.
- Order 2--Placebo Then JNJ Active: Placebo pill used for one week quit attempt, as part of crossover design, followed by one week of trying to quit on active JNJ drug.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week.
  Placebo pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week.
Period: Drug Condition 1: First Study Phase
Arm/Group | Order 1--JNJ Active Then Plac | Order 2--Placebo Then JNJ Active
Started | 18 | 18
Completed | 17 | 15
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3
Period: Drug Condition 2: Second Study Phase
Arm/Group | Order 1--JNJ Active Then Plac | Order 2--Placebo Then JNJ Active
Started | 17 | 15
Completed | 17 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Healthy smokers interested in permanently quitting smoking within the next few months.
Groups:
- Order 1--JNJ Active Then Plac: 200 mg (100 mg b.i.d.) Active JNJ Drug used to assess quitting for one week, as part of crossover design, then one week trying to quit on placebo. This JNJ experimental compound has NO name, just a company number.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week.
  Placebo pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week.
- Order 2--Placebo Then JNJ Active: Placebo pill used for one week quit attempt, as part of crossover design, then one week trying to quit on active JNJ drug.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week.
  Placebo pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week.
- Total: Total of all reporting groups
Arm/Group | Order 1--JNJ Active Then Plac | Order 2--Placebo Then JNJ Active | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36
Fagerstrom Test of Nicotine Dependence (FTND) scale score [Mean (Standard Deviation); unit: units on a scale] — All completed the Fagerstrom Test of Nicotine Dependence (FTND) scale score at baseline, to assess severity of current nicotine dependence. FTND scores range from 0-10, and higher scores index more severe dependence. These scores were not used to determine eligibility, just to characterize dependence severity.
  units on a scale | 4.9 (1.5) | 4.9 (1.5) | 4.9 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Quit Status
Description: Complete abstinence from smoking for 24 hr is counted as a "quit day" and is assessed daily from Mon-Fri for just one week, on the JNJ active drug and one week on placebo. This same Mon-Fri procedure for one week (only) is done for both drug phases. Total outcome in each drug condition therefore is number of quit days out of the five assessment days (range 0-5).
Time Frame: up to one week each drug phase (0-5)
Population: Smokers trying to quit each day during 5-day period on active JNJ, and then during 5-day period on placebo, in crossover design.
Measure: Mean (Standard Deviation); unit: number of days quit
Groups:
- Order 1--JNJ Active Then Plac: 200 mg (100 mg b.i.d.) Active JNJ Drug used to assess quitting for one week, as part of crossover design, then one week quitting on placebo. This JNJ experimental compound has NO name, just a company number.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week.
  Placebo pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week.
- Order 2--Placebo Then JNJ Active: Placebo pill used for one week quit attempt, as part of crossover design, then one week quitting on active JNJ drug.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week.
  Placebo pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week.
Arm/Group | Order 1--JNJ Active Then Plac | Order 2--Placebo Then JNJ Active
Number analyzed (Participants) | 17 | 14
number of days quit
  on JNJ | 0.5 (1.3) | 0.2 (0.6)
  on placebo | 0.7 (1.5) | 0.5 (1.0)

2. Secondary Outcome: Minnesota Nicotine Withdrawal Scale (MNWS) During Attempt to Quit on Active JNJ Drug and on Placebo
Description: Severity of withdrawal symptoms will be assessed with standard self-report measure of Minnesota Nicotine Withdrawal Scale (MNWS) each quit day during one week only on active JNJ, and each quit day during one week on placebo. Ratings are made on 0-100 visual analog scale, with 0="not at all" to 100="very much", and are averaged to create a total score also ranging from 0-100. Higher scores indicate more severe withdrawal.
Time Frame: only on days quit while on JNJ or on placebo
Population: Withdrawal severity on quit days for smokers interested in quitting soon, while attempting to quit briefly during one week on active JNJ or one week on placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Order 1--JNJ Active Then Plac | Order 2--Placebo Then JNJ Active
Number analyzed (Participants) | 17 | 14
units on a scale
  on active JNJ | 12.4 (8.1) | 24.0 (23.4)
  on placebo | 15.5 (15.2) | 23.1 (19.8)

3. Secondary Outcome: Cognitive Function on Continuous Performance Task (CPT) for Those With CO<10 During First Assessment Day (Mon) of Attempt to Quit Smoking During Both JNJ and Plac Quit Periods
Description: This measure of cognitive performance (mean of median speed of correct responding on computer keyboard to letters and numbers) was assessed only on Monday (day 1) of the 0-5 days during each drug/placebo condition. Data only from those shown to have CO<10 ppm were analyzed, to confirm responding during abstinence while on drug/placebo condition. Cognitive testing consisted of standard Continuous Performance Task (CPT), on active JNJ and on placebo phases. This measure is assessed to determine potential mechanism of drug efficacy in relieving disrupted cognitive processing function caused by tobacco deprivation and withdrawal.
Time Frame: first day during quit week on JNJ, and during quit week on placebo.
Population: Only those participants able to quit or sharply limit smoking exposure during both JNJ and the placebo phases of testing, defined as those with CO<10 during both tests of cognitive performance when tobacco abstinent.
Measure: Mean (Standard Deviation); unit: ms time of correct responding
Arm/Group | Order 1--JNJ Active Then Plac | Order 2--Placebo Then JNJ Active
Number analyzed (Participants) | 6 | 6
ms time of correct responding
  on active JNJ | 444.3 (69.3) | 443.3 (32.0)
  on placebo | 434.2 (33.5) | 439.2 (28.0)

ADVERSE EVENTS:
Time Frame: Assessed over the 2 weeks of med use on each condition (active JNJ, or placebo) per participant and ending within 1 week post-participation.
Description: Participants were asked about any adverse effects during each visit. If they reported any, study staff probed for details and contacted study physician who oversaw physical exam at screening to discuss next steps - e.g. monitor and further follow up visits until resolved, or refer to other medical specialists, or to WPIC laboratory for further testing until resolved. Participants also received lab tests via blood sample and EKG at one visit during each 2-week med use period.
Groups:
- While on Active JNJ: 200 mg (100 mg b.i.d.) Active JNJ Drug used to assess quitting for one week, as part of crossover design, followed by one week of quitting on placebo. This JNJ experimental compound has NO name, just a company number.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug used for one week while attempting to briefly quit smoking on Mon-Fri of that week.
- While on Placebo: Placebo pill used for one week quit attempt, as part of crossover design, followed by one week of quitting on active JNJ drug.
  Placebo pill: Placebo pill taken daily to assess ability to briefly quit smoking on Mon-Fri for one week.
Arm/Group | While on Active JNJ | While on Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 5/36 | 3/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | While on Active JNJ (N=36) | While on Placebo (N=36)
self-reported nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) — Self-report of nausea
Abnormal EKG (Cardiac disorders) | 1 (1) | 0 (0) — sinus bradycardia, incomplete right bundle branch QRS pattern
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Self-reported complaint of diahrrea
self-reported skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Skin rash report
swelling in feet (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — swelling, numbness, and pain in feet while walking
body aches (General disorders) | 1 (1) | 0 (0) — Self-reported body aches
feeling of subjective panic (General disorders) | 1 (1) | 1 (1) — Shortness of breath, dizziness, overwhelming feeling
heart racing (Cardiac disorders) | 0 (0) | 1 (1) — heart racing, sadness

LIMITATIONS AND CAVEATS:
Our findings could be specific to the brief duration, procedures used, and single dose tested in this cross-over study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02217527/Prot_SAP_000.pdf